CLINICAL TRIAL: NCT01337843
Title: Wellness Workbook: Efficacy of an Online CBT Workbook for Chronic Low Back Pain
Brief Title: Online Cognitive Behavioral Therapy (CBT) Workbook
Acronym: WW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talaria, Inc (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AR052569; 5R44AR052569-03 (NIH)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; cognitive behavioral pain management; coping; mindfulness; physical activity; Back Pain Lower Back Chronic
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Control Group participants will receive a well-regarded book for back pain patients.
  Interventions: Other: Pain Management Print Materials
- Wellnes Workbook (Experimental): Participants will receive the Wellness Workbook, a web-based cognitive behavioral pain management intervention to help individuals with chronic low back pain (CLBP) learn adaptive coping and pain management skills, increase their physical activity and manage stress with relaxation and mindfulness training
  Interventions: Other: Wellness Workbook

INTERVENTIONS:
Other: Wellness Workbook — A web-based cognitive behavioral pain management intervention to help individuals with chronic low back pain (CLBP) learn adaptive coping and pain management skills, increase physical activity and manage stress. This is a 10 week intervention. Participants use one chapter of the workbook each week. Each chapter takes approximately 1.5 hours to complete.
  Arms: Wellnes Workbook
Other: Pain Management Print Materials — Print materials comparable to the content within Wellness Workbook
  Arms: Control Group

SUMMARY:
This research will evaluate the efficacy of a new online self- help intervention, the Wellness Workbook, for individuals with chronic low back pain (CLBP). Participants will be randomly assigned to use the Wellness Workbook or alternative self-help materials and assessed at baseline, post-intervention (10 weeks) and at follow-up (18 weeks). Outcome measures include pain-related disability and pain severity.

DETAILED DESCRIPTION:
This research will evaluate the efficacy of a new online self- help intervention, the Wellness Workbook, for individuals with chronic low back pain (CLBP). The Wellness Workbook is an interactive online intervention that uses evidence-based cognitive behavioral therapy (CBT) strategies, behavioral activation and mindfulness training to increase chronic pain patients' quality of life. 198 patients with chronic low back pain will be randomly assigned to use the Wellness Workbook or alternative self-help materials for 10 weeks. Participants will be assessed at baseline, post-intervention (10 weeks) and at follow-up (18 weeks). Outcome measures include pain-related disability, pain severity, physical activity, mindfulness and pain-related attitudes and beliefs.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing chronic non-cancer pain in the lower back

Exclusion Criteria:

* has a health diagnosis that would prevent him/her from participating fully in the program (e.g., is receiving treatment for cancer)
* does not have regular Internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Lower pain related disability and interference scores. | Baseline, 10 weeks, 18 weeks
  As compared to the control group participants, CLBP patients who use the WW intervention will report lower pain-related disability and lower pain interference scores.

SECONDARY OUTCOMES:
Fewer pain-related disabling beliefs and attitudes. | Baseline, 10 weeks, 18 weeks
  As compared to the control group participants, CLBP patients who use the WW will report fewer pain-related disabling beliefs and attitudes, have better self-efficacy for managing pain and negative affect and will score higher on mindfulness/present moment awareness. They will also have higher physical activity scores and lower depression scores.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stoner, Ph.D., Principal Investigator — Talaria, Inc
Locations (1):
- Talaria Inc, Seattle, Washington, United States